CLINICAL TRIAL: NCT06666660
Title: Centrum; the Effect of Daily Intake of Multivitamin & Mineral Supplementation, on Biological Age in Relatively Healthy Middle-aged Individuals (CEDIRA)
Brief Title: Daily Intake of Multivitamin & Mineral Supplementation Effects on Biological Age of Relatively Healthy Middle-aged Individuals
Acronym: CEDIRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: HALEON (Industry)
Responsible Party: Principal Investigator, Andrea Maier, Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CEDIRA-NUS; HALEON (Other Grant/Funding Number: HALEON)
Record Dates: First submitted 2024-10-23; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Relatively Healthy Volunteers
Keywords: multivitamin; supplement; randomized controlled trial; biological age; DNA methylation; Epigenetic age
MeSH Terms: interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multivitamin/Mineral Supplement (MVM) (Experimental): Participants in this arm will take 1.2g/day of MVM supplement from CENTRUM for 12 months.
  Interventions: Dietary Supplement: Multivitamin/Mineral supplements
- Placebo (Placebo Comparator): Participants in this arm will take 1.2g/day of placebo for 12 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Multivitamin/Mineral supplements — Each participant will be given 180 MVM tablets in bottles at baseline visit, and another 180 tablets at 6-month visit. Participants will be advised to take 1 tablet orally daily, in the morning before food. Participants will be asked to return the remainder of dispensed MVM tablets, along with the bottle when they come for visit 2 and visit 3. This is done for investigational product accounting and checking for adherence to the assigned treatment arm.
  Arms: Multivitamin/Mineral Supplement (MVM)
Other: Placebo — Each participant will be given 180 placebo tablets in bottles at baseline visit, and another 180 tablets at 6-month visit. Participants will be advised to take 1 tablet orally, daily, in the morning before food. Participants will be asked to return the remainder of dispensed placebo tablets, along with the bottle when they come for visit 2 and visit 3. This is done for investigational product accounting and checking for adherence to the assigned treatment arm. The placebo pills and bottles will be identical in appearance as MVM to ensure effective blinding.
  Arms: Placebo

SUMMARY:
Micronutrients, such as vitamins and minerals, are required to sustain fundamental physiological processes in individuals. As individuals age, the risk of having suboptimal levels of micronutrients increases due to several age-related changes affecting their digestion and assimilation processes. Suboptimal levels of micronutrients have been associated with increased risk of chronic diseases and accelerated ageing. Three years intake of a multivitamin and mineral supplement (MVM) improved global cognition, episodic memory and executive function in older adults. Furthermore, suboptimal micronutrient levels have been associated with a higher biological age, and diet and lifestyle interventions might lower the biological age measured by methylation clocks. Therefore, further evaluation is warranted to determine if MVM supplementation could improve the biological age and clinical outcomes in individuals with a higher biological age.

DETAILED DESCRIPTION:
Accelerated ageing, characterized by a reduced function of multiple organ systems, can be measured by biological, clinical and digital biomarkers of aging. These biomarkers of aging are used to express the biological age of individuals. A higher biological age is not only associated with suboptimal micronutrients levels, but can also be reduced through lifestyle intervention, dietary intervention and nutrient supplementation. A frequently used biological biomarker of ageing is DNA methylation (DNAm) status, which is measured using a set of algorithm known as DNAm clock. This value has been accepted as a good indicator to capture fundamental molecular processes tied to the ageing process. Several studies using Vitamin D, Vitamin B12, and Vitamin C and E have shown positively modify DNAm clock, thus biological age. Henceforth, this study aims to determine if MVM supplementation can reduce the biological age in participants who are biologically older as assessed by DNAm clock.

Rationale for Study Population Middle aged individuals with a high biological age have a high risk of age-releated disesases. Efforts are being made to prevent the development and incidence of age-related diseases and therewith to reduce healthcare costs. Relatively healthy (no chronic disease), middle-aged (40-60 (inclusive) years old) individuals with a biological age higher than their chronological age will be included in this randomized, double-blinded, placebo-controlled trial.

Rationale for Study Design CEDIRA is a randomized, double-blinded, placebo-controlled trial including relatively healthy middle-aged individuals with a higher biological age to evaluate the effect of MVM supplementation for 12 months on biological age and other clinical and biological characteristics such as micronutrient levels in blood, anthropometrics, glucose control, lipid profile, cognition, muscle strength, skin health, lifestyle behaviour, and quality of life.

ELIGIBILITY:
Inclusion Criteria

Participants will be recruited if they fall in the following categories:

1. Relatively healthy middle aged (40-60 years) man or woman;
2. Completed the pre-screening requirements and has managed to schedule the screening visit;
3. Met the randomization criteria after the screening visit i.e., your biological age (as measured by blood DNA methylation) is greater than the chronological age;
4. Able to attend all 4 research visits for screening and research data collection at the NUHS Centre for Healthy Longevity (CHL) at Alexandra Hospital or MD11, National University of Singapore.
5. Willing to wear an OURA ring for 14 consecutive days after each study visits.
6. Willing to download study platform application into their mobile phone throughout the study period.

Exclusion Criteria

Participants will NOT be recruited if they fall in any one or more of the following categories:

1. BMI lower than 18 kg/m2 or higher than or equal to 30 kg/m2 [25];
2. Pre-existing, or history of major cardiovascular diseases (coronary artery disease, heart failure, stroke, peripheral vascular disease, pulmonary hypertension), severe/uncontrolled hypertension (more than 1 prescribed medication), rheumatic heart disease, congenital heart disease, deep vein thrombosis, pulmonary embolism;
3. Type 1 diabetes and Type 2 diabetes;
4. Active cancer or treatment of cancer in the last 3 years;
5. Chronic obstructive pulmonary disease (COPD), severe asthma (taking daily medications);
6. Pregnant women or women planning pregnancy in the next 12 months;
7. Multiple sclerosis or autoimmune/immune deficiency diseases such as Rheumatic arthritis, HIV, Crohn's disease;
8. Recent history of sepsis or infection (within 3 months of in-patient hospitalisation);
9. Any psychiatric disease or neurodegenerative diseases such as Alzheimer's Disease, Parkinson's Disease, Lewy body dementia, and any eating disorders;
10. Hepatitis and liver cirrhosis (independent of severity);
11. Severe kidney disease (GFR less than 30 ml/min/1.73 m2);
12. Skin disease (on systemic medication);
13. Individuals who are on another trial that requires them taking similar or partially similar investigational product (Appendix 1);
14. Individuals who are advised by their medical practitioner to take a MVM supplement;
15. Refuse to stop taking any non-prescribed supplements that contain the investigational product (Appendix 1) within one month before the screening visit and during the study period;
16. Taking a medically prescribed supplements that contains 2 or more of the ingredients of the investigational product (Appendix 1);
17. Individuals with planned hospitalization in the next 12 months;
18. Any serious medical illness which in the PI's judgment may jeopardise the participant by his or her participation in this study or may hamper his or her ability to perform and complete procedures required in the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in blood DNA methylation status, years | Baseline, 6 months and 12 months
  DNA methylation aging clock

SECONDARY OUTCOMES:
Body Mass Index (BMI) change | Baseline, 6 months and 12 months
  comparison of BMI at baseline, interim and end of trial
Waist-to-hip ratio change | Baseline, 6 months and 12 months
  comparison of waist-to-hip ratio at baseline, interim and end of trial
Body fat mass (kg) change | Baseline, 6 months and 12 months
  comparison of body fat mass at baseline, interim and end of trial
Skeletal muscle mass (kg) change | Baseline, 6 months and 12 months
  comparison of skeletal muscle mass at baseline, interim and end of trial
Percentage body fat (%) change | Baseline, 6 months and 12 months
  comparison of percentage body fat at baseline, interim and end of trial
Systolic blood pressure (mm Hg) change | Baseline, 6 months and 12 months
  comparison of systolic blood pressure at baseline, interim and end of trial
Diastolic blood pressure (mm Hg) change | Baseline, 6 months and 12 months
  comparison of diastolic blood pressure at baseline, interim and end of trial
Pulse rate (BPM) change | Baseline, 6 months and 12 months
  comparison of pulse rate at baseline, interim and end of trial
Skin elasticity (mm/time) change | Baseline, 6 months and 12 months
  comparison of skin elasticity measured by he resistance of the skin to the negative pressure (firmness) and its ability to return into its original position (elasticity) displayed as curves (penetration depth in mm/time) at baseline, interim and end of trial
Skin colour (L* a* b*) change | Baseline, 6 months and 12 months
  comparison of skin colour measured using automatic calculation of ITA (Individual Typology Angle) that uses CIE L* a* b* values to classify 6 skin colours from very light to dark at baseline, interim and end of trial
Skin autofluorescence (au) change | Baseline, 6 months and 12 months
  comparison of skin autofluorescence levels calculated by dividing the mean value of the emitted light intensity per nm between 420 and 600 nm by the mean value of the excitation light intensity per nm between 300 and 420 nm, expressed in arbitrary units (AU) at baseline, interim and end of trial
Complete blood count | Baseline, 6 months and 12 months
  comparison of blood count at baseline, interim and end-of-trial
Change in immune parameters: complete blood count | Baseline, 6 months and 12 months
  comparison of immune parameters at baseline, interim and end-of-trial.
Change in immune parameters: inflammatory parameters in serum (mg/dL) | Baseline, 6 months, 12 months
  comparison of immune parameters at baseline, interim and end-of-trial
Change in clinical blood parameters: renal function (mg/dL) | Baseline, 6 months and 12 months
  comparison of clinical blood parameters at baseline, interim and end-of-trial
Change in clinical blood parameters: lipid profile test (mmol/L) | Baseline, 6 months and 12 months
  comparison of clinical blood parameters at baseline, interim and end-of-trial
Change in clinical blood parameters: glucose (mg/dL) | Baseline, 6 months and 12 months
  comparison of clinical blood parameters at baseline, 6 months and 12 months
Change in clinical blood parameters: insulin (mg/dL) | Baseline, 6 months and 12 months
  comparison of clinical blood parameters at baseline, interim and end of trial
Change in clinical blood parameters: glycelated haemoglobin, HbA1C (mmol/mol) | Baseline, 6 months and 12 months
  comparison of clinical blood parameters at baseline, interim and end of trial
Change in clinical blood parameters: metabolites (mmol/l) | Baseline, 6 months and 12 months
  comparison of clinical blood parameters at baseline, interim and end of trial
Change in micronutrient levels in blood | Baseline, 6 months and 12 months
  comparison of micronutrient levels in blood at baseline, interim and end of trial
Change in micronutrient levels in urine | Baseline, 6 months and 12 months
  comparison of micronutrient levels in urine at baseline, interim and end of trial
Change in cognition (Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Test) | Baseline, 6 months and 12 months
  comparison of cognition at baseline, interim and end of trial
Change in handgrip strength change (kg) | Baseline, 6 months and 12 months
  comparison of handgrip strength at baseline, interim and end of trial
Change in quality of life (EuroQoL-5D-5L) | Baseline, 6 months and 12 months
  comparison of quality of life at baseline, interim and end of trial
Change in sleep quality (modified Pittsburgh Sleep Quality Questionnaire) | Baseline, 6 months and 12 months
  comparison of sleep quality at baseline, interim and end of trial
Change in sleep quality (Satisfaction, Alertness, Timing, Efficiency and Duration (SATED) Questionnaire) | Baseline, 6 months and 12 months
  comparison of sleep quality at baseline, interim and end of trial
Change in dietary intake (3-day Food Record) | Baseline, 6 months and 12 months
  comparison of dietary intake at baseline, interim and end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Britta Maier, MD PhD FRACP, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - Healthy Longevity Translational Research Programme, Level 3, MD 11, 10 Medical Dr, Yong Loo Lin School of Medicine, National University of Singapore, Singapore, Singapore
  - Center for Healthy Longevity, Clinic L, Alexandra Hospital, 378 Alexandra Road, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No